CLINICAL TRIAL: NCT01298674
Title: Epidemiological Study of the Prevalence of Age-Related Macular Degeneration in Portugal
Status: Completed | Type: Observational
Sponsor: Association for Innovation and Biomedical Research on Light and Image (Other)
Responsible Party: Sponsor
Other Study IDs: CC-01-2009
Record Dates: First submitted 2011-02-15; First posted 2011-02-18 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an epidemiological study to assess the the prevalence of Age-Related Macular (ARM) Degeneration in Portugal.

ELIGIBILITY:
Inclusion Criteria:

* Participants with 55 years-old

Exclusion Criteria:

* None

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with 55 or more years-old
Sampling Method: Probability Sample
Enrollment: 6023 (Actual)
Dates: Start 2009-08; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
ARM | 1 month after the screening
  Signs of Age-Related Macular Degeneration

SECONDARY OUTCOMES:
Other ocular disease | 1 month after screening
  Signs of other ocular disease such as: diabetic retinopathy, glaucoma, cataract, etc.

CONTACTS AND LOCATIONS:
Overall Officials: José Cunha-Vaz, MD, PhD, Study Director — Association for Innovation and Biomedical Research on Light and Image; Rufino Silva, MD, PhD, Principal Investigator — Association for Innovation and Biomedical Research on Light and Image
Locations (2):
- Portugal (2):
  - Health care units of Lousã and Trevim-Sol, Lousã, Coimbra District
  - ARS Centro - Centro de Saúde de Mira, Mira